CLINICAL TRIAL: NCT03010215
Title: Treatment of Chronic Diabetic Foot Ulcers by Minimally Invasive Surgery in a Cross-sectional Study
Brief Title: Treatment of Chronic Diabetic Foot Ulcers by Minimally Invasive Surgery
Acronym: DiabeticMIS1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Carlo Biz, MD, Assistant Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DiabeticMIS01
Record Dates: First submitted 2016-12-20; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Diabetic Foot Infection; Diabetic Foot Ulcer Neuropathic; Deformities Foot
Keywords: Minimally Invasive Surgery; Percutaneous distal osteotomy; Distal Metatarsal Minimally-invasive Osteotomy (DMMO); Percutaneous Tenotomy; Forefoot; Metatarsal bones
MeSH Terms: conditions — Diabetic Foot; Foot Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minimally Invasive Surgery (MIS) (Other): Patients with plantar chronic diabetic foot ulcers will be treated by Distal Metatarsal Minimally invasive Osteotomy (DMMO).
  Interventions: Other: Distal Metatarsal Minimally invasive Osteotomy (DMMO)

INTERVENTIONS:
Other: Distal Metatarsal Minimally invasive Osteotomy (DMMO) — Percutaneous dorsal incision at the level of the the distal part of the metatarsal bone, a Shannon burr is introduced at the level of metatarsal neck, with orientation of at approximately 45°, keeping the articular cartilage surface of the metatarsal head as reference point on the superior cortex.
  In this position, under fluoroscopic control, the osteotomy is started following a distal-dorsal and proximal-plantar direction. In this way the metatarsal head moves proximally and dorsally reducing the metatarsal pressure on the plantar ulcer.

SUMMARY:
Despite the development of the control of DM and the great interest for the complications of the disease, even today the diabetic foot represents a challenge for the orthopaedic surgeon. Being frequently correlated to alteration of the plantar pressures, the surgery treatment is recommended and the Minimally Invasive Surgery (MIS) candidates itself to solve this pathologic case.

The purpose of this longitudinal cross-sectional study was to evaluate radiographic and surgical outcomes and the subjective grade of satisfaction of the patients with a diagnosis of chronic plantar diabetic foot ulcers that have been treated at Padua's Orthopaedic Clinic through MIS.

DETAILED DESCRIPTION:
Thirty-two patients with chronic diabetic foot ulcers (CDFUs) were treated by MIS between January 2010 and September 2016. Clinical evaluation was assessed pre-operatively, as well as at 3 months after surgery and at final follow-up, using the American Orthopaedic Foot and Ankle Society (AOFAS) Hallux Metatarsophalangeal-Interphalangeal Scale. The recurrence of the ulcers and complications were recorded. All the ulcers were evaluated with the University of Texas Diabetic Wound Classification. We used the radiological Maestro's criteria to evaluated the radiographs before and after the operation. Also, the bridging bone/callus formation was evaluated at the different radiographic follow-ups, while the articular surface congruency. The global disability was evaluated with the Short Form Health Survey (SF-36) and the satisfaction's level with the Visual Analogue Scale (VAS). Statistical analysis was carried out using the Wilcoxon signed-rank test. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM;
* presence of a plantar CDFU, so not healed after 6 months of medical multidisciplinary treatment;
* HbA1c < 8,5%.

Exclusion Criteria:

* congenital deformities of the foot;
* macroscopic signs of local infection of the soft tissues;
* alteration of CRP>150 mg/L;
* previous foot and ankle surgery;
* previous foot and ankle surgery;
* rheumatic, neurologic, infective, or psychiatric pathologies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2016-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Score change of the AOFAS Hallux metatarsophalangeal interphalangeal scale | From 1 month before the operation until study completion, an average of 2 years.
  Total between 0 to 100.

SECONDARY OUTCOMES:
Radiological outcomes changes after surgical treatment | Preoperative and at 3-6-12 months post-operative
  Evaluation of the Maestro Criteria and the bridging bone/callus formation.
Change in clinical evaluation with SF-36 score | From 1 month before the operation until study completion, an average of 2 years.
Change in clinical evaluation with VAS | From 1 month before the operation until study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Biz, MD, Principal Investigator — University of Padova
Locations (1):
- Orthopaedic Clinic, Padua University, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Yes
Age, Gender, Radiological and Clinica parameters and images.

REFERENCES:
- [Result] Biz C, Fosser M, Dalmau-Pastor M, Corradin M, Roda MG, Aldegheri R, Ruggieri P. Functional and radiographic outcomes of hallux valgus correction by mini-invasive surgery with Reverdin-Isham and Akin percutaneous osteotomies: a longitudinal prospective study with a 48-month follow-up. J Orthop Surg Res. 2016 Dec 5;11(1):157. doi: 10.1186/s13018-016-0491-x. PMID 27919259
- [Result] Tamir E, Finestone AS, Avisar E, Agar G. Mini-Invasive floating metatarsal osteotomy for resistant or recurrent neuropathic plantar metatarsal head ulcers. J Orthop Surg Res. 2016 Jul 11;11(1):78. doi: 10.1186/s13018-016-0414-x. PMID 27401772
- [Result] Dayer R, Assal M. Chronic diabetic ulcers under the first metatarsal head treated by staged tendon balancing: a prospective cohort study. J Bone Joint Surg Br. 2009 Apr;91(4):487-93. doi: 10.1302/0301-620X.91B4.21598. PMID 19336809
- [Result] Henry J, Besse JL, Fessy MH; AFCP. Distal osteotomy of the lateral metatarsals: a series of 72 cases comparing the Weil osteotomy and the DMMO percutaneous osteotomy. Orthop Traumatol Surg Res. 2011 Oct;97(6 Suppl):S57-65. doi: 10.1016/j.otsr.2011.07.003. Epub 2011 Aug 27. PMID 21873138